CLINICAL TRIAL: NCT03821389
Title: Airway Clearance Using Non-Invasive Oscillating Device in Critically Ill Children
Brief Title: Airway Clearance Using Non-Invasive Oscillating Device
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: MedTeq (Industry)
Responsible Party: Principal Investigator, Atsushi Kawaguchi, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000
Record Dates: First submitted 2019-01-17; First posted 2019-01-29 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Insufficiency
Keywords: Chest Physiotherapy; Non-invasive; Oscillation; Secretion
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIOD Frequencer of 40Hz (Experimental): 40 Hz of NIOD will be applied and then 60Hz will be used 3 hours later. 60 Hz of NIOD will be applied and then 40Hz will be used 3 hours later for the rest of the patients. The investigators will analyze the difference in average effects between 40Hz and 60Hz.
  Interventions: Device: NIOD Frequencer
- NIOD Frequencer of 60Hz (Active Comparator)
  Interventions: Device: NIOD Frequencer

INTERVENTIONS:
Device: NIOD Frequencer — NIOD will be implemented on four different parts of the chest walls, 3 minutes for each part and 12 minutes in total per each session. Left and right front and posterior chest walls will be stimulated (Figure1), particularly, on the anterior chest, intercostal spaces 1-2 above nipple line and lateral side of the midclavicular line 1-2 below intercostal spaces. The intensity of the NIOD can be selected between 80-100%, which is prespecified on the machine.

SUMMARY:
This study aims to examine the tolerance, feasibility, and physiological effects in airway clearance by using a novel non-invasive oscillating transducer device (NIOD, FrequencerTM) in critically ill children. The project is two years long with two separate stages of investigation. This study specifically examines different frequencies of NIOD to find the best frequency on patients outcomes.

DETAILED DESCRIPTION:
Airway obstruction due to excessive production of secretion in small children especially those with bronchiolitis is a critical problem in the clinical management. Chest physiotherapy (CPT) and an invasive positive percussion ventilation (IPPV) have been recognized as to encourage dislodging the secretions; nonetheless, the tolerance to the procedure and its efficiency have not been proved to be sufficient. This study aims to examine the tolerance, feasibility, and physiological effects in airway clearance by using a novel non-invasive oscillating transducer device (NIOD) in critically ill children. The study will be prospective Crossover Randomized Study in a Pediatric Intensive Care Unit in a Canadian Academic Children's Hospital. We will target children less than 24-month-old, for whom CPT is prescribed for airway clearance with or without atelectasis. We will apply two different frequencies of NIOD (i.e. 40 and 60Hz) for 3 minutes each, on each patient 3 hours apart. The investigators will apply a pragmatic design, so that other procedures including hypertonic saline nebulization, IPPV, suctioning (e.g., oral or nasal), or changing the ventilator settings or modality (i.e., increasing PEEP or changing the nasal mask to total face CPAP) can be provided at the direction of bedside pediatric intensivists in charge.

ELIGIBILITY:
Inclusion Criteria:

* All the patients admitted to the PICU during the study period will be screened. The investigators will not set any restriction regarding the timing of prescription of CPT (i.e., length of PICU stay before screening) for the screening. The investigators will include only if CPT is expected to be used as a management at least for the next 24 hours in the PICU from the time of inclusion. For instance, if CPT will be expected to be discontinued from the management in a day, the investigators will exclude the participants from the inclusion. CPT can be prescribed for airway clearance with any etiology such as atelectasis at the directions of bedside pediatric intensivists in charge on the study date. The investigators will only include patients whose oxygenation is stable (SpO2>90%) with less than 0.60 of ventilators.

Exclusion Criteria:

* CPT order will (or is expected to) be discontinued within 24 hours from the inclusion timing.
* CPT is not ordered for airway clearance.
* SpO2 is not stable (SpO2=<90%) with more than 0.60 of FIO2 for the ventilated patients including patients on NIV, at least for previous 1 hour from the screening.
* SpO2 is not stable (SpO2=<90%) with more than 0.60 of FIO2 for the patients on HFNC, at least for previous 1 hour from the screening.
* Bradycardia (HR<80bpm) at any interventions at least for 24 hours prior to the screening.
* Patients with known pneumothorax, osteomyelitis in the PICU admission.
* Known pulmonary hypertension with treatment(s) underway.
* Thoracotomy within 1 month.
* Known recent/unhealed rib fractures.
* Known skin injury of chest wall.
* No obtain of IC.
* Brain death or vegetated states.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean changes in respiratory tidal volume | 1) right before the intervention being initiated, 2) right after the end of the intervention (i.e., 12 minutes from 1)), and 3) 30 min after each intervention finished.
  Tidal volume will be measured by non-invasive 3D system for non-intubated patients and ventilator for intubated patients.

SECONDARY OUTCOMES:
Changes of blood pressures (mmHg) | from the beginning of the intervention till 30 min after the intervention will be extracted from the Electronic Medical Records (i.e., every minutes).
Estimated lung volume | 1) right before the intervention being initiated, 2) right after the end of the intervention (i.e., 12 minutes from 1)), and 3) 30 min after each intervention finished.
  lung volume will be measured by mechanical ventilator when patients are on an invasive mechanical ventilator, or 3D non-invasive measuring system when patients are not on an invasive mechanical ventilator (reference: Computerized Medical Imaging and Graphics 70 (2018) 17-28)
EtCO2 and its waveform. | Baseline: before the procedure, Comparison: two minutes from the beginning of the procedure
Clinical Respiratory severity scores | collected 1) right before the intervention being initiated, 2) right after the end of the intervention (i.e., 12 minutes from 1)), and 3) 30 min after each intervention finished.
  Use modified Woods Score, which consists of 5 elements including 1) accessory muscle use 2) cyanosis (Y/N), 3) lung air entry, 4) level of contiousness, and 5) wheeze (Y/N). The score scales from 0-10, for which the higher score indicates higher severity of respiratory condition.
Change of heart rates (beat per minute) | from the beginning of the intervention till 30 min after the intervention will be extracted from the Electronic Medical Records (i.e., every minutes).
Change of oxygen saturations (%) | from the beginning of the intervention till 30 min after the intervention will be extracted from the Electronic Medical Records (i.e., every minutes).
Change of respiratory rate (times per minute) | from the beginning of the intervention till 30 min after the intervention will be extracted from the Electronic Medical Records (i.e., every minutes).
Change of neurological status (i.e., patient comfort level). | 1) right before the intervention being initiated, 2) right after the end of the intervention (i.e., 12 minutes from 1)), and 3) 30 min after each intervention finished.
  Use COMFORT-B Scale. Score scale: 1-35, higher scale indicates that patients is more agitated and uncomfortable.
Change of level of work of breathing (i.e., no WOB, mild, moderate, and severe). | 1) right before the intervention being initiated, 2) right after the end of the intervention (i.e., 12 minutes from 1)), and 3) 30 min after each intervention finished.
Lung air distribution | 1) right before the intervention being initiated, 2) right after the end of the intervention (i.e., 12 minutes from 1)), and 3) 30 min after each intervention finished.
  lung air distribution will be measured by using EIT (electrical impedance tomography). The distribution will be examined by area of air distribution which is measured and quantified by EIT.

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Kawaguchi, Principal Investigator — St. Justine's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kawaguchi A, Bernier G, Adler A, Emeriaud G, Jouvet PA. Incremental effect of non-invasive oscillating device on chest physiotherapy in critically ill children: a cross-over randomised trial. BMJ Open. 2020 Oct 5;10(10):e038648. doi: 10.1136/bmjopen-2020-038648. PMID 33020101